CLINICAL TRIAL: NCT03316508
Title: Copeptin- Relevance as a Perioperative Marker in Pediatric Cardiac Surgery
Status: Completed | Type: Observational
Sponsor: Claudia Herbst (Other)
Responsible Party: Sponsor-Investigator, Claudia Herbst, Dr. med. univ., Medical University of Vienna
Organization: Medical University of Vienna (Other)
Other Study IDs: CHS1706001
Record Dates: First submitted 2017-10-02; First posted 2017-10-20 (Actual); Last update posted 2019-09-11 (Actual); Status verified 2019-09

CONDITIONS: Congenital Heart Disease
Keywords: copeptin; pediatric cardiac surgery; heart lung machine
MeSH Terms: conditions — Heart Defects, Congenital; Diabetes Insipidus

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — EDTA blood samples
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This study evaluates the relevance of Copeptin in children with congenital heart disease undergoing cardiac surgery with the need of cardiopulmonary bypass. Three blood samples are taken of each patient. The first and second sample are collected in the operation room before and after the procedure and the third sample on the first postoperative day at the intensive care unit.

DETAILED DESCRIPTION:
Objective:

Vasopressin is a hormone secreted by the posterior pituitary gland. Its main functions are constriction of blood vessels and reabsorption of water and thereby regulating water balance and hemodynamics of the body. Copeptin is a cleavage product in the synthesis of vasopressin and is released in equimolar amounts. Its stability makes it easier to determine the amount of vasopressin. It is known, that the use of a heart-lung machine in cardiac procedures has effects on the water balance of the body and may affect the vasopressin secretion.

The aim of this prospective clinical trial is, to figure out if copeptin would be suitable for perioperative risk evaluation in neonates and children with congenital heart disease after surgery with the use of a heart-lung machine.

Hypotheses:

The primary outcome endpoint of this study is the change in copeptin concentration perioperatively in patients with congenital heart disease, with the use of heart-lung machine.

Secondary outcome endpoints are correlations between copeptin concentration and complexity of the procedure (based on the aristotle basic score), clinical status and the perfusion times of the heart-lung machine.

ELIGIBILITY:
Inclusion Criteria:

* ≤6 years of age
* CHD
* need of HLM for surgery
* Informed consent of parents
* not participating in other studies

Exclusion Criteria:

* Preoperative ventilatory support
* Preoperative circulatory support (ECMO, VAD)
* Diabetes insipidus
* Preoperative CPR
* Preoperative shock
* Preoperative sepsis
* Preoperative vasopressin application

Max Age: 6 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: The study population consists of 81 patients (neonates, infants, children) with congenital heart disease and the need of cardiac surgery with a heart-lung machine. Parental consent after pre-operative consultation and informing about the study is required.
Sampling Method: Non-Probability Sample
Enrollment: 81 (Actual)
Dates: Start 2017-06-14 (Actual); Primary Completion 2018-10-01 (Actual); Study Completion 2019-08-10 (Actual)

PRIMARY OUTCOMES:
Change of Copeptin concentrations | baseline and up to one day
  Change of Copeptin concentrations between the baseline and first postoperative measurement

SECONDARY OUTCOMES:
Intubation | up to one day
  Duration of intubation time
Cardiopulmonary bypass | up to one day
  Total time of cardiopulmonary bypass and aortic cross clamp time.
ICU stay | up to one day
  Length of ICU stay
Complexity of procedures | up to one day
  The surgical complexity of the procedures undergone by the patients will be shown by using a scoring system developed for this purpose named Aristotle Score

CONTACTS AND LOCATIONS:
Overall Officials: Claudia R Herbst, MD, Principal Investigator — Medical University Vienna Department for Cardiac Surgery
Locations (1):
- Medical University of Vienna, Vienna, Austria

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2017-04-17): https://cdn.clinicaltrials.gov/large-docs/08/NCT03316508/Prot_SAP_000.pdf
  • Informed Consent Form (2017-04-27): https://cdn.clinicaltrials.gov/large-docs/08/NCT03316508/ICF_001.pdf